CLINICAL TRIAL: NCT03033719
Title: Multicenter Randomized Trial Comparing Laparoscopy and Laparotomy for Colon Cancer Surgery in Patients Older Than 75 Years
Brief Title: Colectomy for Cancer in the Elderly by Laparoscopy or Laparotomy
Acronym: CELL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K130901; 2016-A00312-49 (Other: ID RCB)
Record Dates: First submitted 2017-01-10; First posted 2017-01-27 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Colonic Cancer
Keywords: Colorectal Surgery; Geriatrics; Digestive Oncology; Colon cancer; Elderly patients; Laparoscopy; Laparotomy; Morbidity
MeSH Terms: conditions — Colonic Neoplasms | interventions — Laparotomy; Conversion to Open Surgery; Laparoscopy; Minimally Invasive Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparotomy (Active Comparator): Open surgery
  Interventions: Procedure: Laparotomy
- Laparoscopy (Experimental): Minimally invasive surgery
  Interventions: Procedure: Laparoscopy

INTERVENTIONS:
Procedure: Laparotomy — Open surgery
  Other Names: Open surgery
  Arms: Laparotomy
Procedure: Laparoscopy — Minimally invasive surgery
  Other Names: Minimally invasive surgery
  Arms: Laparoscopy

SUMMARY:
The purpose of this study is to compare the postoperative global morbidity between patients who have been operated on for a colon cancer by laparotomy and those operated on by laparoscopy

DETAILED DESCRIPTION:
The present study is a national, multicenter, open-label randomized, 2-arm superiority trial. Patients aged 75 years or older with uncomplicated colonic cancer or precancerous colonic lesion non-endoscopically resectable, will be randomized to either colectomy by laparoscopy or laparotomy. All patients that might be included will have a comprehensive geriatric assessment performed within the 30 days before randomization with the following scores: MMS (Mini Mental Score), ADL scale (Activities of Daily Living), IADL scale (Instrumental Activities of Daily Living), GDS (Geriatric Depression Scale) and TGUG test ("Timed Get-Up-and-Go" test).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 75 years
2. Histologically proven colonic adenocarcinoma (> 15 cm from the anal margin) or precancerous colonic lesion non endoscopically resectable
3. Uncomplicated colonic tumor (no preoperative suspicion of invasion of adjacent structures as assessed by CT-scan (cT4), no tumoral perforation, or tumoral obstruction, or abscess, or hemorrhage)
4. No previous colonic cancer within the 5 last years
5. No peritoneal carcinosis on CT-scan
6. Patient able to fill in an auto-questionnaire alone or with some help
7. MMS (Mini Mental Score) ≥ 15
8. Given oral consent (formal informed consent is not required by French law for accepted procedures)

Exclusion Criteria:

1. Rectal cancer (≤ 15 cm from the anal margin)
2. Locally advanced (cT4) or complicated tumor requiring extended resection or emergency surgery
3. Synchronous colonic cancer
4. - Scheduled need for synchronous intra-abdominal surgery, including surgery for liver metastases
5. Absolute contraindications to general anesthesia or prolonged pneumoperitoneum
6. Patient not able to tolerate colon surgery according to the global comprehensive geriatric assessment
7. Estimated life expectancy less than 6 months
8. Patient under guardianship
9. Other known active cancer (except nonmelanomatous skin cancer)
10. Patient not affiliated to the social security system
11. Previous colonic resection

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2017-07-04 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Global postoperative morbidity in both arms | At 30 days after the surgery
  Postoperative morbidity is defined as any surgical or medical complications occurring up to 30 days after surgery. It will be collected using a standardized collection form during hospitalization and eventual subsequent consultations in case of patient discharge before then

SECONDARY OUTCOMES:
Postoperative mortality | Evaluated at 30 days and at 90 days after the surgery
  Death from any cause
Rate of readmission | Within the 30 days after discharge of the patient
  Defined as any rehospitalization whatever the cause
Number of examined lymph nodes | At surgery
  Quality of surgical resection : Number of examined lymph nodes
Type of resection (R0 or R1) | At surgery
  Quality of surgical resection : Type of resection (R0 or R1)
Pathological evaluation of mesocolic resection quality | At surgery
  Quality of surgical resection : Pathological evaluation of mesocolic resection quality
Health-related quality of life : Quality of Life Questionnaires (EORTC QLQ-C30) | At randomization and three months postoperatively
  Health-related quality of life : Quality of Life Questionnaires (EORTC QLQ-C30)
Health-related quality of life : Quality of Life Questionnaires (EORTC QLQ-CR29) | At randomization and three months postoperatively
  Health-related quality of life : Quality of Life Questionnaires (EORTC QLQ-CR29)
Mini Mental State (MMS) Examination or Folstein test | Before randomization and three months postoperatively
  Evolution of geriatric scores : The Mini Mental State (MMS) Examination or Folstein test; (Comprehensive geriatric assessment performed by a geriatrician on each site)
Katz Activities of Daily Living (ADL) scale | Before randomization and three months postoperatively
  Evolution of geriatric scores :The Katz Activities of Daily Living (ADL) scale (Comprehensive geriatric assessment performed by a geriatrician on each site)
Geriatric Depression Scale (GDS) | Before randomization and three months postoperatively
  Evolution of geriatric scores :The Geriatric Depression Scale (GDS) (Comprehensive geriatric assessment performed by a geriatrician on each site)
Timed Get-up-and-go (TGUG) | Before randomization and three months postoperatively
  Evolution of geriatric scores :The Timed Get-up-and-go (TGUG) test (Comprehensive geriatric assessment performed by a geriatrician on each site)

OTHER OUTCOMES:
To establish a specific molecular classification of colon cancer in the elderly from expression chips | within the 15 years after the tumor sampling
  To establish a specific molecular classification of colon cancer in the elderly from expression chips (Ancillary studies will be conducted from formalin fixed paraffin embedded (FFPE) tumor samples from our cohort)
To establish associations between molecular subtypes, the clinical and histological factors and relevant genetic alterations | within the 15 years after the tumor sampling
  To establish associations between molecular subtypes, the clinical and histological factors and relevant genetic alterations (Ancillary studies will be conducted from formalin fixed paraffin embedded (FFPE) tumor samples from our cohort)
To establish a possible link between these molecular subtypes and overall survival of patients | within the 15 years after the tumor sampling
  To establish a possible link between these molecular subtypes and overall survival of patients.
  (Ancillary studies will be conducted from formalin fixed paraffin embedded (FFPE) tumor samples from our cohort)
To compare our molecular classification with the different classifications already published in the literature on colorectal cance | within the 15 years after the tumor sampling
  To compare our molecular classification with the different classifications already published in the literature on colorectal cancer (Ancillary studies will be conducted from formalin fixed paraffin embedded (FFPE) tumor samples from our cohort)

CONTACTS AND LOCATIONS:
Overall Officials: Gilles MANCEAU, M.D., PhD.,, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Groupe Hospitalier Pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Manceau G, Brouquet A, Chaibi P, Passot G, Bouche O, Mathonnet M, Regimbeau JM, Lo Dico R, Lefevre JH, Peschaud F, Facy O, Volpin E, Chouillard E, Beyert-Berjot L, Verny M, Karoui M, Benoist S. Multicenter phase III randomized trial comparing laparoscopy and laparotomy for colon cancer surgery in patients older than 75 years: the CELL study, a Federation de Recherche en Chirurgie (FRENCH) trial. BMC Cancer. 2019 Dec 4;19(1):1185. doi: 10.1186/s12885-019-6376-8. PMID 31801485